CLINICAL TRIAL: NCT05401838
Title: Piloting a Brief Cognitive-Behavioral Therapy (BCBT) Group Intervention for Suicidal Behavior Among Active Duty Military Personnel
Brief Title: The Group Risk Reduction Intervention Therapy (GRRIT) Project
Acronym: ProjectGRRIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Collaborators: Ohio State University (Other); United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert J. Cramer, PhD, Belk Endowed Professor in Health Research, University of North Carolina, Charlotte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH2210234; CDMRP-PR210136 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-05-24; First posted 2022-06-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Suicidal Ideation; Suicide, Attempted; Coping Skills; Depression; Anxiety; PTSD
Keywords: Randomized controlled trial; Group therapy; Military
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Investigators will conduct parallel 2-arm randomized controlled trial of G-BCBT compared to a DBT skills group. G-BCBT is a new adaptation of the existing BCBT protocol administered in a group format. Because DBT's efficacy in a group format is already supported and investigators anticipate G-BCBT to be at least as equally effective, investigators propose a 2-arm non-inferiority design.
Who Masked: Outcomes Assessor
Masking Description: Co-I Gunn (statistician) will be blinded to intervention condition during primary data analyses; the dataset will be cleaned by other project staff and intervention condition will be referred to only as intervention A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-BCBT (Experimental): 68 active duty service member participants assigned to G-BCBT will undergo 12 group therapy sessions scheduled on a weekly basis.
  Interventions: Behavioral: Group Brief Cognitive-Behavioral Therapy (G-BCBT)
- DBT (Active Comparator): 68 active duty service member participants in the DBT condition will receive 24 weekly group therapy sessions each lasting 90 minutes.
  Interventions: Behavioral: Dialectical Behavior Therapy (DBT) Skills Group

INTERVENTIONS:
Behavioral: Group Brief Cognitive-Behavioral Therapy (G-BCBT) — G-BCBT comprises 12, 90 minute sessions organized in three phases: (1) emotion regulation, (2) cognitive flexibility, and (3) relapse prevention. The first session will be a tailored individual session focusing on person-specific crisis response planning and developing the participant's suicide mode. Sessions 2 through 5 feature treatment goal setting, followed by teaching skills in stimulus control, mindfulness, relaxation, a reasons for living task, and survival kit. Sessions 6 through 10 provide opportunities for improving cognitive flexibility via cognitive-behavioral exercises such as ABC worksheets, challenging questions, patterns of problematic thinking worksheets, coping cards, and activity planning. The third phase of treatment focuses on relapse prevention, and encompasses the last two sessions of treatments where group participants demonstrate mastery of the skills learned in treatment and practice successfully navigating a future stressful situation.
  Arms: G-BCBT
Behavioral: Dialectical Behavior Therapy (DBT) Skills Group — DBT comprises 24 weekly group therapy sessions each lasting 90 minutes. DBT sessions include worksheets and skills practice activities. The DBT protocol entails three phases as follows. Phase I (8 weeks) covers a two-week mindfulness orientation and a six-week distress tolerance module. Distress tolerance skill building includes paired muscle relaxation, distraction, and radical acceptance. Phase II (nine weeks) entails a two-week mindfulness module followed by seven weeks of emotion regulation skill building. Emotion regulation content includes a model of describing emotion and a pleasant events checklist. Phase III (7 weeks) includes two-week mindfulness and orientation module, followed by five weeks of interpersonal effectiveness training. Interpersonal effectiveness training approaches include clarifying goals in interpersonal situations, guidelines for keeping relationships, and self-respect. Mindfulness, cutting across modules, addresses review of concepts such as Wise Mind.
  Arms: DBT

SUMMARY:
Investigators will evaluate a group format adaptation of Brief Cognitive-Behavioral Therapy for Suicide (i.e., G-BCBT) on suicide ideation (Aim 1), ability to use coping strategies (Aim 2), and overall mental health (exploratory analysis). The combination of tailored means safety counseling and training in evidence-based emotion regulation and cognitive flexibility skills delivered via a 12-session group therapy treatment will decrease service members' overall suicide risk. The group format will provide opportunities to learn and practice skills, thereby enhancing self-efficacy. G-BCBT outcomes are expected to be no worse than Dialectical Behavior Therapy (DBT) group skills training, an existing gold standard intervention that is twice the length of time as G-BCBT.

DETAILED DESCRIPTION:
Background: The suicide rate among active duty service members is more than double the civilian population in the United States. Also, approximately 1 in 20 service members report suicidal ideation each year, and 1 in 100 service members report a non-fatal suicide attempt annually. Suicidal behavior rates are compounded by a number of mental health services access barriers such as clinician shortages. The purpose of this randomized controlled trial (RCT) is to demonstrate that a new group therapy intervention protocol, Group Brief Cognitive-Behavioral Therapy (G-BCBT) for Suicide, will positively impact suicidal behavior, mental health, and self-regulatory skill outcomes for service members experiencing recent suicidal behavior.

Hypotheses/Objectives: The overall objective of the proposal is to evaluate the effects of a G-BCBT protocol on suicidal ideation, suicide attempts, mental health, and self-regulatory skills. Investigators expect that G-BCBT will result in improved service member suicidal behavior (Aim 1), ability to use coping strategies (Aim 2), and overall mental health (exploratory analysis). The combination of tailored means safety counseling and training in evidence-based emotion regulation and cognitive flexibility skills will improve service members' self-control. The group format will provide opportunities to learn and practice skills, thereby enhancing self-efficacy. G-BCBT outcomes are expected to be no worse than Dialectical Behavior Therapy (DBT) group skills training, an existing gold standard intervention that is twice the length of time as G-BCBT. Secondary hypotheses are that G-BCBT will (a) demonstrate non-inferior improvements in self-regulatory skills, and (b) self-regulatory skills will moderate G-BCBT's impact on suicidal ideation.

Specific Aims: Investigators expect this project will yield mental health and coping skills benefits for service members. These expected outcomes will be attained through the following aims: Aim 1: Pilot a group format of BCBT for its impact on suicidal behavior among active duty military service members; Aim 2: Assess the relationship between G-BCBT and self-regulatory factors.

Study Design: This study employs a single-site 4-year, 2-arm phase III RCT design. Data will be collected at Naval Medical Center Portsmouth. University of North Carolina at Charlotte will coordinate the study and conduct intervention evaluation. The Ohio State University will conduct fidelity monitoring and provide treatment subject matter expertise for both conditions. A total of 136 active duty service members will be randomly assigned to one of two conditions: (1) G-BCBT or (2) DBT. Service members in the G-BCBT condition will complete a 12-week protocol comprising tailored means safety counseling followed by emotion regulation and cognitive flexibility skills training. Service members assigned to the DBT condition will complete a 24-week protocol covering mindfulness, emotion regulation, distress tolerance, and interpersonal effectiveness skills training. All participants will complete assessments at baseline, after each session, upon treatment completion, and 3- and 6-months post-intervention completion. Data will address suicidal behavior, mental health, self-regulatory skills, treatment process factors, and demographic and suicide-related covariates.

Clinical Impact: G-BCBT will be tested as an evidence-based suicide-specific intervention requiring less resources compared to available options. This study will result in the following knowledge products that will be distributed to military healthcare system and community stakeholders: G-BCBT protocol, revised BCBT manual, train-the-trainer materials, technical report, suicide prevention white paper, and G-BCBT fidelity assessment materials. This study supports in the 2015 Department of Defense (DoD) Strategy for Suicide Prevention and 2019 Veterans Affairs/DoD Clinical Practice Guidelines for the Assessment and Management of Patients at Risk for Suicide. G-BCBT lethal means counseling and coping skills training will enhance service member quality of life and operational readiness.

This randomized controlled clinical trial will test a new suicide-specific group therapy intervention, Group-Brief Cognitive-Behavioral Therapy for Suicide (G-BCBT), by comparing it to an established gold standard.

ELIGIBILITY:
Inclusion Criteria:

* (1) Be an active duty service member.
* (2) Be 18 years-of-age or older.
* (3) Be of treatment-seeking status in outpatient mental health or substance abuse rehabilitation clinics, and/or inpatient psychiatry discharge.
* (4) Report current suicide ideation within the last week and/or a suicide attempt within the past month.
* (5) Be able to understand and speak English.
* (6) Possess ability to complete the informed consent process.

Exclusion Criteria:

* (1) Have a psychiatric or medical condition that precludes the ability to provide informed consent or participation in outpatient treatment (e.g., psychosis, mania, acute intoxication).
* (2) Retired service members and family/dependents.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Scale for Suicidal Ideation score | From pre-intervention baseline to 3- and 6-months post-treatment completion.
  Suicidal ideation will be measured with the Beck Scale for Suicide Ideation (BSSI). The BSSI contains 19 self-report items assessing of suicidal ideation. With a score range of 0 to 38, higher scores reflect worse ideation. The BSSI demonstrates strong reliability and associations with suicide measures when used with military personnel.

SECONDARY OUTCOMES:
Frequency of suicide attempts | From pre-intervention baseline to 3- and 6-months post-treatment completion.
  Suicide attempts will be defined as intentional self-injurious behavior for which there is evidence of intent to die. We will measure suicide attempts using the Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R), a structured clinician-administered interview that assesses features of suicide attempts and other self-injurious behaviors. The SITBI-R will be converted to self-report format. The full version will be administered at baseline. Only the suicide attempt question will be administered at follow-up time-points. Also, question time frames will be reworded to reflect last point of contact (e.g., since last therapy session). The SITBI-R has demonstrated good construct validity. Review of the U.S. military's Behavioral Health Data Portal (BHDP) medical records will additionally be conducted to identify suicide attempts that might have been missed during SITBI-R administrations (e.g., participants who drop out early or miss follow-up assessments).
Change in Patient Health Questionnaire-9 score | From pre-intervention baseline to 3- and 6-months post-treatment completion.
  Depression will be quantified with the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 contains nine self-report items measuring of depression symptom severity. With a score range of 0 to 27, higher scores reflect worse depressive symptoms. The PHQ-9 has demonstrated high internal consistency among treatment-seeking service members, and construct validity in a clinical sample.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Cramer, PhD, Principal Investigator — UNC Charlotte
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual datasets with de-identified complete data with data dictionaries will be available; however, interested parties will need to request specific variables via completion of a Data Request Form (DSF). The DSF contains requestor name, position, affiliation, contact information, summary of research questions and aims, description of the data/code to be requested, an anticipated project timeline, and study team, roles and authorship list for the proposed project. The DSF will be reviewed by the Project Investigator Committee, comprising PI Cramer, Co-PI Baker, Co-Bryan, Co-I Gunn, and Co-I Franks. To be granted, the DSF must (a) be determined to not overlap with study team project aims, or current/planned analyses, and (b) be accepted by majority vote in writing. If the request is denied or deemed pending revision, PI Cramer or Co-PI Baker will provide the requestor a signed copy of the DSF with a short explanation of the determination.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available 6 months after the end of the project grant period. Data and supplemental materials identified above will be available in perpetuity.
Access Criteria: See above (Data Request Form).

REFERENCES:
- [Result] Rudd MD, Bryan CJ, Wertenberger EG, Peterson AL, Young-McCaughan S, Mintz J, Williams SR, Arne KA, Breitbach J, Delano K, Wilkinson E, Bruce TO. Brief cognitive-behavioral therapy effects on post-treatment suicide attempts in a military sample: results of a randomized clinical trial with 2-year follow-up. Am J Psychiatry. 2015 May;172(5):441-9. doi: 10.1176/appi.ajp.2014.14070843. Epub 2015 Feb 13. PMID 25677353
- [Result] Cramer RJ, Franks M, Cunningham CA, Bryan CJ. Preferences in Information Processing: Understanding Suicidal Thoughts and Behaviors among Active Duty Military Service Members. Arch Suicide Res. 2022 Jan-Mar;26(1):169-186. doi: 10.1080/13811118.2020.1760156. Epub 2020 May 5. PMID 32369420
- [Derived] Baker JC, Grover S, Gunn LH, Charles C, Rikli H, Franks MJ, Khazem LR, Williams S, Ammendola E, Washington C, Bennette M, Starkey A, Schnecke K, Cain S, Bryan CJ, Cramer RJ. Group brief cognitive behavioral therapy for suicide prevention compared to dialectal behavior therapy skills group for military service members: a study protocol of a randomized controlled trial. BMC Psychiatry. 2023 Dec 5;23(1):904. doi: 10.1186/s12888-023-05282-x. PMID 38053122

DOCUMENTS (1):
  • Informed Consent Form (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT05401838/ICF_002.pdf